CLINICAL TRIAL: NCT02682446
Title: Prediction for the Development of Metachronous Gastric Cancer After Endoscopic Submucosal Dissection by Serum Pepsinogen
Brief Title: The Efficacy of Serum Pepsinogen for Prediction of Metachronous Gastric Neoplasm
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Seong Woo Jeon, Professor, Kyungpook National University Hospital
Other Study IDs: KNUMC_13-1059
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Cancer
Keywords: Early gastric cancer; endoscopic submucosal dissection; serum pepsinogen; Helicobacter pylori
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum pepsinogen, serum HP IgG
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Negative H. pylori group: The participants revealed negative findings of H pylori IgG and other invasive methods (rapid urease test or histology) at the time of ESD for EGC
- Previous H. pylori infection group: The participants revealed positive findings of H pylori IgG and other invasive methods (rapid urease test or histology) at the time of ESD for EGC
- Eradicated H. pylori group: The participants revealed to success for H. pylori eradication in those who were positive findings of H pylori IgG and other invasive methods (rapid urease test or histology) at the time of ESD for EGC
  Interventions: Drug: H pylori eradication
- Persistent H. pylori group: The participants revealed to fail in H. pylori eradication in those who were positive findings of H pylori IgG and other invasive methods (rapid urease test or histology) at the time of ESD for EGC
  Interventions: Drug: H pylori eradication

INTERVENTIONS:
Drug: H pylori eradication — The regimen of H. pylori eradication was like that: 1-week conventional proton pump inhibitor (PPI) based triple therapy (lansoprazole 40 mg b.i.d., clarithromycin 500 mg b.i.d., and amoxicillin 1 g b.i.d. for a week) after confirmation of H. pylori infection. If the participants who initially failed to respond to the first eradication, they recommended to underwent second-line eradication therapy with the regimen of 7-day bismuth containing quadruple regimen [lansoprazole 40 mg b.i.d., tripotassium dicitrate bismuthate (Denol; Greencross Co., Seoul, Korea) 300 mg q.i.d. (three tablets 30 min before meals and one tablet 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d. for 1 week]
  Groups: Eradicated H. pylori group; Persistent H. pylori group

SUMMARY:
After endoscopic resection of early gastric cancer (EGC), there remained concerned about the development of the metachronous gastric neoplasm (MGN). The aim of this study was to evaluate the role of H. pylori eradication for reducing MGN after ESD and the efficacy of serum pepsinogen (PG) for predicting development of MGN after endoscopic submucosal dissection (ESD) for EGC and to evaluate other risk factors for the incidence of MGN. The investigators enrolled the participants who were tested serum PG I and II at the time of ESD for EGC, from January 2007 to May 2013 in single tertiary center, retrospectively. The baseline characteristics of the participants, H. pylori status, and serum pepsinogen were analyzed for the development of the MGN.

ELIGIBILITY:
Inclusion Criteria:

* The patients who tested serum PG concentration test and H. pylori status at the time of ESD and revealed pathologically complete en bloc resection after ESD for EGC.

Exclusion Criteria:

* previous history of ER; proven pathologically incomplete resection or lympho-vascular invasion on the resected ESD specimen; additional treatment after ESD; and follow-up loss less than 2 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was designed to enroll patients in our ESD data registry, prospectively. Finally, we analyzed the data retrospectively. We enrolled about more than 1000 patients in our ESD registry. For this cohort study, we enrolled about 800 patients for analysis.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2007-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence (number of participants) of metachronous gastric neoplasm after ESD between H. pylori eradicated group and H. pylori persistent group | Up to 8 years after ESD for EGC
  The investigators were estimated the number of participants who found metachronous gastric neoplasm after ESD for EGC during follow up endoscopic surveillance. Then, the investigator will evaluate the statitistical difference in the incidence of the development of metachornous gastric neoplasm between H. pylori eradicated group and H. pylori persistent group.

SECONDARY OUTCOMES:
To evaluate the incidence of metachronous gastric neoplasm after ESD based on diffferent cut off point of serum pepsinogen. | Up to 8 years after ESD for EGC
  The investigators will evaluate the incidence of metachronous gastric neoplasm after ESD using several cut off level of serum pepsinogen: 30, 50 and 70 ng/mL for PG I and 3 for PG I/II ratio. The appropriate cut off level could be found for indicating the development of metachronous gastric neoplasm using serum PG

CONTACTS AND LOCATIONS:
Overall Officials: Seong Woo Jeon, Prof., Principal Investigator — Gastric cancer center, Kyungpook national university medical center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fukase K, Kato M, Kikuchi S, Inoue K, Uemura N, Okamoto S, Terao S, Amagai K, Hayashi S, Asaka M; Japan Gast Study Group. Effect of eradication of Helicobacter pylori on incidence of metachronous gastric carcinoma after endoscopic resection of early gastric cancer: an open-label, randomised controlled trial. Lancet. 2008 Aug 2;372(9636):392-7. doi: 10.1016/S0140-6736(08)61159-9. PMID 18675689
- [Result] Abe S, Oda I, Suzuki H, Nonaka S, Yoshinaga S, Nakajima T, Sekiguchi M, Mori G, Taniguchi H, Sekine S, Katai H, Saito Y. Long-term surveillance and treatment outcomes of metachronous gastric cancer occurring after curative endoscopic submucosal dissection. Endoscopy. 2015 Dec;47(12):1113-8. doi: 10.1055/s-0034-1392484. Epub 2015 Jul 10. PMID 26165734
- [Result] Choi KS, Jung HY, Choi KD, Lee GH, Song HJ, Kim DH, Lee JH, Kim MY, Kim BS, Oh ST, Yook JH, Jang SJ, Yun SC, Kim SO, Kim JH. EMR versus gastrectomy for intramucosal gastric cancer: comparison of long-term outcomes. Gastrointest Endosc. 2011 May;73(5):942-8. doi: 10.1016/j.gie.2010.12.032. Epub 2011 Mar 9. PMID 21392757
- [Result] Suzuki R, Yamamoto E, Nojima M, Maruyama R, Yamano HO, Yoshikawa K, Kimura T, Harada T, Ashida M, Niinuma T, Sato A, Nosho K, Yamamoto H, Kai M, Sugai T, Imai K, Suzuki H, Shinomura Y. Aberrant methylation of microRNA-34b/c is a predictive marker of metachronous gastric cancer risk. J Gastroenterol. 2014 Jul;49(7):1135-44. doi: 10.1007/s00535-013-0861-7. Epub 2013 Aug 13. PMID 23942619
- [Result] Bae SE, Jung HY, Kang J, Park YS, Baek S, Jung JH, Choi JY, Kim MY, Ahn JY, Choi KS, Kim DH, Lee JH, Choi KD, Song HJ, Lee GH, Kim JH. Effect of Helicobacter pylori eradication on metachronous recurrence after endoscopic resection of gastric neoplasm. Am J Gastroenterol. 2014 Jan;109(1):60-7. doi: 10.1038/ajg.2013.404. Epub 2013 Dec 17. PMID 24343545
- [Result] Samloff IM, Varis K, Ihamaki T, Siurala M, Rotter JI. Relationships among serum pepsinogen I, serum pepsinogen II, and gastric mucosal histology. A study in relatives of patients with pernicious anemia. Gastroenterology. 1982 Jul;83(1 Pt 2):204-9. No abstract available. PMID 7084603
- [Result] Watabe H, Mitsushima T, Yamaji Y, Okamoto M, Wada R, Kokubo T, Doi H, Yoshida H, Kawabe T, Omata M. Predicting the development of gastric cancer from combining Helicobacter pylori antibodies and serum pepsinogen status: a prospective endoscopic cohort study. Gut. 2005 Jun;54(6):764-8. doi: 10.1136/gut.2004.055400. PMID 15888780
- [Derived] Kwon Y, Jeon S, Nam S, Shin I. Helicobacter pylori infection and serum level of pepsinogen are associated with the risk of metachronous gastric neoplasm after endoscopic resection. Aliment Pharmacol Ther. 2017 Oct;46(8):758-767. doi: 10.1111/apt.14263. Epub 2017 Aug 11. PMID 28799258